CLINICAL TRIAL: NCT00972010
Title: A Prospective, Controlled Study To Evaluate Surgical Excision Margins in Malignant Breast Lumpectomies With the PEAK PlasmaBlade Compared to Traditional Electrosurgery
Brief Title: Study to Evaluate Surgical Excision Margins in Malignant Breast Lumpectomies With the PEAK PlasmaBlade
Status: Completed | Type: Observational
Sponsor: Sarah Blair, M.D. (Other)
Collaborators: Medtronic Surgical Technologies (Industry)
Responsible Party: Sponsor-Investigator, Sarah Blair, M.D., Professor of Surgery, University of California, San Diego
Organization: University of California, San Diego (Other)
Other Study IDs: 090314
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
Keywords: Breast; Cancer; Lumpectomies; PlasmaBlade; Breast conservation therapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Breast tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to find out more about distinguishing between cancerous and non-cancerous breast cancer cells at the edges of tumors. Using an FDA approved device to remove tumors, this device will be tested to see if it causes less tissue damage and therefore makes it easier to examine the tumor and make sure it is all excised. The tumors will be excised by standard surgical technique, and then the effects of the device on the removed tissues will be studied.

DETAILED DESCRIPTION:
Breast conservation therapy (BCT) is the standard surgical treatment for breast cancer. The goal of BCT is total excision of the malignant lesion while simultaneously preserving the cosmetic appearance and functionality of the breast. Despite advances in technique and pathologic analysis; however, 20-50% of malignant breast lump excisions have cancer present to the edge of the excision margin (defined as a "positive" margin). Excisions that are found to be margin positive require a secondary excision; however, in these cases residual disease is found to be present in only 40-70% of cases. Some researchers have hypothesized that re-excision was unnecessary in a certain percentage of cases. Currently there are no routinely utilized method for intra-operative interpretation of surgical margins. Touch preps or imprint cytology has been used in the past in some centers but it is not used routinely because an experienced cytopathologist is needed to correctly interpret the slides.

The standard of care to evaluate surgical margins is based on permanent section. Margins are considered negative if there is greater than 1 mm of normal tissue between cancer cells to the excised surface. Many factors for this discrepancy have been postulated, including artifact associated with the inking process and with electrosurgery induced damage of the margin during excision (thermal injury); therefore, creating a "false positive" impression of tumor cells present at surgical margins. We propose a clinical study to evaluate the effects of thermal injury in breast cancer excision using traditional electrosurgery (i.e., the "Bovie") compared to the pulsed RF technology with the PEAK PlasmaBlade. We hypothesize that the PlasmaBlade will impart less thermal injury to the incised breast tissue (malignant and normal) and will increase the specificity of the margin status. The majority of breast cancers are removed by traditional electrocautery. We are just starting to utilize this new technology for soft tissue dissection at UCSD.

The PEAK PlasmaBlade is a family of disposable surgical cutting and coagulation devices that offer the exacting control of a scalpel and the bleeding control of traditional electrosurgery without extensive collateral damage. The PlasmaBlade is based on proprietary pulsed plasma technology. This technology represents an evolutionary leap in the advancement of radiofrequency surgical technologies, which originated with traditional electrosurgery and progressed to plasma-mediated energy devices. The PlasmaBlade tissue dissection devices are FDA-cleared and commercially available.

ELIGIBILITY:
Inclusion Criteria

* Women or men with an established diagnosis of an invasive ductal carcinoma
* Women or men with tumors > 1cm
* Women undergoing Breast Conservation Operations
* Women or men may have had prior chemotherapy as long as their treatment was completed >2 weeks prior to enrollment with recovery from any toxicities

Exclusion Criteria

* No established diagnosis of breast cancer
* Women or men with tumors <1 cm
* Women or men undergoing total mastectomy
* Women or men who have had prior radiation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients recruited from the Moores UCSD Cancer Center and the UCSD Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To compare the thermal injury artifact produced by traditional electrosurgery vs. the PEAK PlasmaBlade by intensive pathologic analysis both by gross inspection, touch imprint, and permanent histologic analysis. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L Blair, MD, Principal Investigator — University of California, San Diego
Locations (3):
- United States (3):
  - Thornton Hospital, La Jolla, California
  - Rebecca and John Moores Cancer Center, La Jolla, California
  - UCSD Medical Center, San Diego, California

REFERENCES:
- [Derived] Ruidiaz ME, Cortes-Mateos MJ, Sandoval S, Martin DT, Wang-Rodriguez J, Hasteh F, Wallace A, Vose JG, Kummel AC, Blair SL. Quantitative comparison of surgical margin histology following excision with traditional electrosurgery and a low-thermal-injury dissection device. J Surg Oncol. 2011 Dec;104(7):746-54. doi: 10.1002/jso.22012. Epub 2011 Jul 8. PMID 21744349